CLINICAL TRIAL: NCT04637399
Title: Circadian Misalignment as a Disease Risk Factor in Inflammatory Bowel Disease
Brief Title: Circadian Misalignment in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16080305
Record Dates: First submitted 2019-08-06; First posted 2020-11-19 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ulcerative Colitis: Participants diagnoses with Ulcerative Colitis.
- Crohn's Disease: Participants diagnosed with Crohn's Disease.

SUMMARY:
This study is to explore the role the sleep/wake cycle (Circadian Rhythm) has on Inflammatory Bowel Disease. Participants will be asked to attend two clinic visits 14 days apart. Participants will complete a packet of questionnaires regarding their health and sleep habits. Over the 14 days between visits participants will be asked to wear a wrist actigraphy device that will measure their sleep-wake activity along with filling in a sleep diary. During the visits, participants will have a physical exam on visit 1 and on visit 2 participants will be asked to give blood, stool, and urine samples. Additionally, participants may also give sigmoid tissue samples during an optional unprepped limited flexible sigmoidoscopy procedure.

DETAILED DESCRIPTION:
The long term goal of this Research proposal is to establish that circadian misalignment is a factor for disease flare in inflammatory bowel disease (IBD). In order to achieve this goal this project will focus on two aspects that are critical to address in the management of IBD - disease course and subclinical inflammation. One of the most challenging aspects of IBD medical care is that IBD has a very heterogeneous disease course. Some patients will quickly progress to surgery despite aggressive medical therapy while others have no disease flares on any medications. In order to address these factors, the investigator will access multiple factors about each IBD patient to determine what their previous disease course has been (history), known factors of their disease that are associated with disease course (location, age of diagnosis, etc), and markers of subclinical inflammation that are established predictors of disease flare. Our overall hypothesis is that circadian misalignment is an important factor in the disease course in IBD. To test this hypothesis, the investigator will conduct a series of experiments in humans to elucidate the role of circadian rhythms in IBD. In Aim 1, the investigator will test the hypothesis that circadian misalignment is present in IBD with an aggressive disease course by analyzing circadian rhythms by wrist actigraphy, urinary melatonin, and chronotype questionnaires. In Aim 2, the investigator will assess markers of subclinical inflammation in the same subjects from Aim1, and analyze established predictors of disease flare such as CRP, intestinal permeability, fecal calprotectin, and mucosal inflammation markers. The goal of this research proposal is to identify whether circadian misalignment is a factor in disease course in IBD. It is not to determine if IBD patients have increased circadian misalignment compared to healthy controls, therefore healthy controls are not used as a comparison group. However, Dr. Burgess and Dr. Levi's labs do have a large historical cohort of over 100 healthy controls that have completed wrist actigraphy measurements and chronotype questionnaires that can be used as a comparison if our hypothesis is proven incorrect.

Experimental Design: Subjects with biopsy proven IBD (N=68) will be recruited, 24 CD (Crohn's Disease) and 24 UC (Ulcerative Colitis). All subjects will be between 18-70 years old. Subjects will be recruited from the Rush University GI Clinic. All subjects will complete questionnaires including IBD demographic history, an IBD quality of life, food timing, sleep questionnaires - PROMIS and RUSATED, and chronotype questionnaires - Owl and Lark and Munich. Each subject will be accessed by the PI for exclusion criteria including: 1) Active IBD (HBI ≥ 5 or Modified HBI ≥5); 2) Major depression (score ≥ 15 or any endorsement of suicidal intent on the Beck Depression; 3) Sleep apnea (score high risk ≥ 2 or more categories on the Berlin Questionnaire)(43); 4) Restless leg syndrome (score ≥ 15 on the IRLS Study Group Rating Scale(44)); 5) Regular use of medications that affect intestinal permeability, and/or endogenous melatonin including metoclopramide, NSAIDs, beta blocker, psychotropic medication, hypnotics and exogenous melatonin products during 4 weeks prior to the study; 6) People who have worked night shifts or crossed more than 2 time zones in the previous month; 7) Any major organ disease - renal impairment (creatinine>1.2 mg/dL - previous EMR labs must be within the past 12 months), diabetes (Hgb-A1c > 6.5% - no history of any form of diabetes); liver disease (LFTs > 1.5x nl - previous EMR labs must be within the past 12 months), or significant cardiac problems; 8) Inability to sign an informed consent.

Subjects that meet these inclusion/exclusion criteria will be assessed by the PI, who will perform a physical exam, take a history, and review prior medical testing. Subjects will matched 1:1 during recruitment so N=12 in both CD and UC with aggressive disease and N=12 in both CD and UC with nonaggressive disease (See Experimental Design). All subjects will then have their sleep patterns recorded by wrist actigraphy (30 sec epochs, Actiwatch Spectrum, Phillips Inc.) for 14 days (±3 days). Wrist actigraphy is a reliable standard means of assessing sleep-wake activity,(45) and will be used to calculate circadian rhythm by dichotomy index and r24. During the 14days (±3 days) subjects will also keep a detailed consensus sleep diary which is a standardized prospective sleep measure.(46) At the end of the 14 days (±3 days), and a day prior to their visit, all subjects will complete an online self-administered 24 hour food recall (ASA24) and 24 h urine collection for urinary melatonin which is also a marker of central circadian rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Age of Diagnosis is < 40 years
* Documented biopsy proven Crohn's Disease or Ulcerative Colitis
* Willing to sign study consent form
* At starting and during the study subject is free of prescription and over the counter medication that can affect melatonin over the past month: over the counter melatonin formulation, NSAID, alpha blocker, beta blocker, calcium channel blocker, benzodiazepine, hypnotic, barbiturate, antiepileptic, antidepressant, antipsychotic, metoclopramide

Exclusion Criteria:

* Active IBD flare (HBI≥5)
* Use of prednisone in the past 4 weeks
* Other forms of colitis, such as indeterminate colitis
* Moderate/severe depression or suicidal thoughts
* Restless leg syndrome
* Sleep apnea
* Surgical history of ileostomy or colectomy with ileal pouch
* Antibiotic use within the last 14 days prior to stool collection
* Active or recent infection in the last 14 days prior to stool collection
* Abnormal bleeding parameters (i.e., prolonged INR), history of easy bruising or bleeding (except rectal bleeding during flare-ups)
* Psychiatric disorder (diagnosis reported or EMR)
* Use of anticoagulants and anti-platelet drugs
* Documented chronic disease (history or current) such as diabetes, lung, heart, eye, autoimmune, seizures, kidney (creatinine >1.2 mg/dL in last 12 months),or liver (AST/ALT >1.5x ULN in last 12 months)
* Night shift work (3 or more nights/week) or more than 2 time zones crossed in past 4 weeks
* Any children <2 years old living at home
* WOMEN ONLY: Currently pregnant
* Non-English speaking
* Participating in other research studies involving research interventions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with Ulcerative Colitis or Crohn's Disease.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Harvey Bradshaw Activity Index | 1 Day
  Disease Activity: Score 0-4
Beck's Depression Index | Past Two Weeks from Date of Visit
  Score: 0-14
International Restless Leg Syndrome Scale | Past Week from Date of Visit
  Score 0-14
Berlin OSA Questionnaire | Past 3 Months
  Meet 0-1 Category
Short Inflammatory Bowel Disease Questionnaire | Past Two Weeks from Date of Visit
  Score: 1-7
Munich Chronotype Questionnaire | Past 3 Months
  Typical Sleep and Wake Habits
Owl and Lark Questionnaire | Past 3 Months
  Extreme morning type 70-86 Moderately morning type 59-69 Neutral type 42-58 Moderately evening type 31-41 Extreme evening type 16-30
ActiWatch | 14 Day Period
  Sleep-Wake Activity Wrist Monitor
Food Timing Questionnaire | 14 Day Period
  Food and Sleep Habit Diary
Sleep Diary | 14 Day Period
  Sleep Record

SECONDARY OUTCOMES:
Urine Samples | 1 Day
  Volume: First 5 hours, Second 19 hours, 24 hours
C-Reactive Protein | 10 Weeks +/- 3 Days
  milligrams per deciliter
Left Sided Colon Tissue Samples | 1 Day
  10 Double Bites with Forceps

CONTACTS AND LOCATIONS:
Overall Officials: Garth Swanson, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Kappelman MD, Rifas-Shiman SL, Porter CQ, Ollendorf DA, Sandler RS, Galanko JA, Finkelstein JA. Direct health care costs of Crohn's disease and ulcerative colitis in US children and adults. Gastroenterology. 2008 Dec;135(6):1907-13. doi: 10.1053/j.gastro.2008.09.012. Epub 2008 Sep 17. PMID 18854185
- [Background] Keefer L, Stepanski EJ, Ranjbaran Z, Benson LM, Keshavarzian A. An initial report of sleep disturbance in inactive inflammatory bowel disease. J Clin Sleep Med. 2006 Oct 15;2(4):409-16. PMID 17557469
- [Background] Ali T, Madhoun MF, Orr WC, Rubin DT. Assessment of the relationship between quality of sleep and disease activity in inflammatory bowel disease patients. Inflamm Bowel Dis. 2013 Oct;19(11):2440-3. doi: 10.1097/MIB.0b013e3182a0ea54. PMID 23945186
- [Background] Singh S, Dera AE, Esteban JPG, Chakradeo PS, Lee AA, Burgess HR, Keshavarzian A, Swanson GR. Tu1992 later chronotype is associated with worse quality of life and biologic use in inflammatory bowel disease. Gastroenterology. 2016; 150(4): S999-S1000.
- [Background] Swanson GR, Gorenz A, Shaikh M, Desai V, Kaminsky T, Van Den Berg J, Murphy T, Raeisi S, Fogg L, Vitaterna MH, Forsyth C, Turek F, Burgess HJ, Keshavarzian A. Night workers with circadian misalignment are susceptible to alcohol-induced intestinal hyperpermeability with social drinking. Am J Physiol Gastrointest Liver Physiol. 2016 Jul 1;311(1):G192-201. doi: 10.1152/ajpgi.00087.2016. Epub 2016 May 19. PMID 27198191
- [Background] Summa KC, Voigt RM, Forsyth CB, Shaikh M, Cavanaugh K, Tang Y, Vitaterna MH, Song S, Turek FW, Keshavarzian A. Disruption of the Circadian Clock in Mice Increases Intestinal Permeability and Promotes Alcohol-Induced Hepatic Pathology and Inflammation. PLoS One. 2013 Jun 18;8(6):e67102. doi: 10.1371/journal.pone.0067102. Print 2013. PMID 23825629
- [Background] Beaugerie L, Sokol H. Clinical, serological and genetic predictors of inflammatory bowel disease course. World J Gastroenterol. 2012 Aug 7;18(29):3806-13. doi: 10.3748/wjg.v18.i29.3806. PMID 22876031
- [Background] Grimstad T, Norheim KB, Isaksen K, Leitao K, Hetta AK, Carlsen A, Karlsen LN, Skoie IM, Goransson L, Harboe E, Aabakken L, Omdal R. Fatigue in Newly Diagnosed Inflammatory Bowel Disease. J Crohns Colitis. 2015 Sep;9(9):725-30. doi: 10.1093/ecco-jcc/jjv091. Epub 2015 May 19. PMID 25994356
- [Background] Ranjbaran Z, Keefer L, Farhadi A, Stepanski E, Sedghi S, Keshavarzian A. Impact of sleep disturbances in inflammatory bowel disease. J Gastroenterol Hepatol. 2007 Nov;22(11):1748-53. doi: 10.1111/j.1440-1746.2006.04820.x. PMID 17914945
- [Background] Shearman LP, Sriram S, Weaver DR, Maywood ES, Chaves I, Zheng B, Kume K, Lee CC, van der Horst GT, Hastings MH, Reppert SM. Interacting molecular loops in the mammalian circadian clock. Science. 2000 May 12;288(5468):1013-9. doi: 10.1126/science.288.5468.1013. PMID 10807566
- [Background] Nakahata Y, Yoshida M, Takano A, Soma H, Yamamoto T, Yasuda A, Nakatsu T, Takumi T. A direct repeat of E-box-like elements is required for cell-autonomous circadian rhythm of clock genes. BMC Mol Biol. 2008 Jan 4;9:1. doi: 10.1186/1471-2199-9-1. PMID 18177499
- [Background] Ramsey KM, Yoshino J, Brace CS, Abrassart D, Kobayashi Y, Marcheva B, Hong HK, Chong JL, Buhr ED, Lee C, Takahashi JS, Imai S, Bass J. Circadian clock feedback cycle through NAMPT-mediated NAD+ biosynthesis. Science. 2009 May 1;324(5927):651-4. doi: 10.1126/science.1171641. Epub 2009 Mar 19. PMID 19299583
- [Background] Laposky AD, Bradley MA, Williams DL, Bass J, Turek FW. Sleep-wake regulation is altered in leptin-resistant (db/db) genetically obese and diabetic mice. Am J Physiol Regul Integr Comp Physiol. 2008 Dec;295(6):R2059-66. doi: 10.1152/ajpregu.00026.2008. Epub 2008 Oct 8. PMID 18843095
- [Background] Hoogerwerf WA, Hellmich HL, Cornelissen G, Halberg F, Shahinian VB, Bostwick J, Savidge TC, Cassone VM. Clock gene expression in the murine gastrointestinal tract: endogenous rhythmicity and effects of a feeding regimen. Gastroenterology. 2007 Oct;133(4):1250-60. doi: 10.1053/j.gastro.2007.07.009. Epub 2007 Jul 12. PMID 17919497
- [Background] Bozek K, Relogio A, Kielbasa SM, Heine M, Dame C, Kramer A, Herzel H. Regulation of clock-controlled genes in mammals. PLoS One. 2009;4(3):e4882. doi: 10.1371/journal.pone.0004882. Epub 2009 Mar 16. PMID 19287494
- [Background] Panda S, Antoch MP, Miller BH, Su AI, Schook AB, Straume M, Schultz PG, Kay SA, Takahashi JS, Hogenesch JB. Coordinated transcription of key pathways in the mouse by the circadian clock. Cell. 2002 May 3;109(3):307-20. doi: 10.1016/s0092-8674(02)00722-5. PMID 12015981
- [Background] Turek FW. Circadian clocks: tips from the tip of the iceberg. Nature. 2008 Dec 18;456(7224):881-3. doi: 10.1038/456881a. No abstract available. PMID 19092918
- [Background] Bell-Pedersen D, Cassone VM, Earnest DJ, Golden SS, Hardin PE, Thomas TL, Zoran MJ. Circadian rhythms from multiple oscillators: lessons from diverse organisms. Nat Rev Genet. 2005 Jul;6(7):544-56. doi: 10.1038/nrg1633. PMID 15951747
- [Background] Ueda HR, Hayashi S, Chen W, Sano M, Machida M, Shigeyoshi Y, Iino M, Hashimoto S. System-level identification of transcriptional circuits underlying mammalian circadian clocks. Nat Genet. 2005 Feb;37(2):187-92. doi: 10.1038/ng1504. Epub 2005 Jan 23. PMID 15665827
- [Background] Nojkov B, Rubenstein JH, Chey WD, Hoogerwerf WA. The impact of rotating shift work on the prevalence of irritable bowel syndrome in nurses. Am J Gastroenterol. 2010 Apr;105(4):842-7. doi: 10.1038/ajg.2010.48. Epub 2010 Feb 16. PMID 20160712
- [Background] Brzozowski T, Zwirska-Korczala K, Konturek PC, Konturek SJ, Sliwowski Z, Pawlik M, Kwiecien S, Drozdowicz D, Mazurkiewicz-Janik M, Bielanski W, Pawlik WW. Role of circadian rhythm and endogenous melatonin in pathogenesis of acute gastric bleeding erosions induced by stress. J Physiol Pharmacol. 2007 Dec;58 Suppl 6:53-64. PMID 18212400
- [Background] Kolstad HA. Nightshift work and risk of breast cancer and other cancers--a critical review of the epidemiologic evidence. Scand J Work Environ Health. 2008 Feb;34(1):5-22. doi: 10.5271/sjweh.1194. PMID 18427694
- [Background] Wong PM, Hasler BP, Kamarck TW, Muldoon MF, Manuck SB. Social Jetlag, Chronotype, and Cardiometabolic Risk. J Clin Endocrinol Metab. 2015 Dec;100(12):4612-20. doi: 10.1210/jc.2015-2923. Epub 2015 Nov 18. PMID 26580236
- [Background] Mazzoccoli G, Palmieri O, Corritore G, Latiano T, Bossa F, Scimeca D, Biscaglia G, Valvano MR, D'Inca R, Cucchiara S, Stronati L, Annese V, Andriulli A, Latiano A. Association study of a polymorphism in clock gene PERIOD3 and risk of inflammatory bowel disease. Chronobiol Int. 2012 Oct;29(8):994-1003. doi: 10.3109/07420528.2012.705935. Epub 2012 Aug 10. PMID 22881285
- [Background] Burgess HJ, Swanson GR, Keshavarzian A. Endogenous melatonin profiles in asymptomatic inflammatory bowel disease. Scand J Gastroenterol. 2010 Jun;45(6):759-61. doi: 10.3109/00365521003749818. No abstract available. PMID 20345337
- [Background] Sandborn WJ, Feagan BG, Hanauer SB, Lochs H, Lofberg R, Modigliani R, Present DH, Rutgeerts P, Scholmerich J, Stange EF, Sutherland LR. A review of activity indices and efficacy endpoints for clinical trials of medical therapy in adults with Crohn's disease. Gastroenterology. 2002 Feb;122(2):512-30. doi: 10.1053/gast.2002.31072. No abstract available. PMID 11832465
- [Background] Panaccione R, Ghosh S, Middleton S, Marquez JR, Scott BB, Flint L, van Hoogstraten HJ, Chen AC, Zheng H, Danese S, Rutgeerts P. Combination therapy with infliximab and azathioprine is superior to monotherapy with either agent in ulcerative colitis. Gastroenterology. 2014 Feb;146(2):392-400.e3. doi: 10.1053/j.gastro.2013.10.052. PMID 24512909
- [Background] D'Inca R, Di Leo V, Corrao G, Martines D, D'Odorico A, Mestriner C, Venturi C, Longo G, Sturniolo GC. Intestinal permeability test as a predictor of clinical course in Crohn's disease. Am J Gastroenterol. 1999 Oct;94(10):2956-60. doi: 10.1111/j.1572-0241.1999.01444.x. PMID 10520851
- [Background] Wyatt J, Oberhuber G, Pongratz S, Puspok A, Moser G, Novacek G, Lochs H, Vogelsang H. Increased gastric and intestinal permeability in patients with Crohn's disease. Am J Gastroenterol. 1997 Oct;92(10):1891-6. PMID 9382060
- [Background] Swanson G, Forsyth CB, Tang Y, Shaikh M, Zhang L, Turek FW, Keshavarzian A. Role of intestinal circadian genes in alcohol-induced gut leakiness. Alcohol Clin Exp Res. 2011 Jul;35(7):1305-14. doi: 10.1111/j.1530-0277.2011.01466.x. Epub 2011 Apr 4. PMID 21463335
- [Background] Preuss F, Tang Y, Laposky AD, Arble D, Keshavarzian A, Turek FW. Adverse effects of chronic circadian desynchronization in animals in a "challenging" environment. Am J Physiol Regul Integr Comp Physiol. 2008 Dec;295(6):R2034-40. doi: 10.1152/ajpregu.00118.2008. Epub 2008 Oct 8. PMID 18843092
- [Background] Natale V, Innominato PF, Boreggiani M, Tonetti L, Filardi M, Parganiha A, Fabbri M, Martoni M, Levi F. The difference between in bed and out of bed activity as a behavioral marker of cancer patients: A comparative actigraphic study. Chronobiol Int. 2015;32(7):925-33. doi: 10.3109/07420528.2015.1053909. PMID 26158757
- [Background] Levi F, Dugue PA, Innominato P, Karaboue A, Dispersyn G, Parganiha A, Giacchetti S, Moreau T, Focan C, Waterhouse J, Spiegel D; ARTBC Chronotherapy Group. Wrist actimetry circadian rhythm as a robust predictor of colorectal cancer patients survival. Chronobiol Int. 2014 Oct;31(8):891-900. doi: 10.3109/07420528.2014.924523. Epub 2014 Jun 13. PMID 24927369
- [Background] Keshavarzian A, Holmes EW, Patel M, Iber F, Fields JZ, Pethkar S. Leaky gut in alcoholic cirrhosis: a possible mechanism for alcohol-induced liver damage. Am J Gastroenterol. 1999 Jan;94(1):200-7. doi: 10.1111/j.1572-0241.1999.00797.x. PMID 9934756
- [Background] Banan A, Choudhary S, Zhang Y, Fields JZ, Keshavarzian A. Ethanol-induced barrier dysfunction and its prevention by growth factors in human intestinal monolayers: evidence for oxidative and cytoskeletal mechanisms. J Pharmacol Exp Ther. 1999 Dec;291(3):1075-85. PMID 10565827
- [Background] Banan A, Fields JZ, Decker H, Zhang Y, Keshavarzian A. Nitric oxide and its metabolites mediate ethanol-induced microtubule disruption and intestinal barrier dysfunction. J Pharmacol Exp Ther. 2000 Sep;294(3):997-1008. PMID 10945852
- [Background] Burgess HJ, Eastman CI. The dim light melatonin onset following fixed and free sleep schedules. J Sleep Res. 2005 Sep;14(3):229-37. doi: 10.1111/j.1365-2869.2005.00470.x. PMID 16120097
- [Background] Burgess HJ, Eastman CI. Early versus late bedtimes phase shift the human dim light melatonin rhythm despite a fixed morning lights on time. Neurosci Lett. 2004 Feb 12;356(2):115-8. doi: 10.1016/j.neulet.2003.11.032. PMID 14746877
- [Background] Burgess HJ, Fogg LF. Individual differences in the amount and timing of salivary melatonin secretion. PLoS One. 2008 Aug 26;3(8):e3055. doi: 10.1371/journal.pone.0003055. PMID 18725972
- [Background] Burgess HJ, Eastman CI. Short nights attenuate light-induced circadian phase advances in humans. J Clin Endocrinol Metab. 2005 Aug;90(8):4437-40. doi: 10.1210/jc.2005-0536. Epub 2005 May 10. PMID 15886231
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956
- [Background] Hening WA, Allen RP. Restless legs syndrome (RLS): the continuing development of diagnostic standards and severity measures. Sleep Med. 2003 Mar;4(2):95-7. doi: 10.1016/s1389-9457(03)00009-1. No abstract available. PMID 14592339
- [Background] de Souza L, Benedito-Silva AA, Pires ML, Poyares D, Tufik S, Calil HM. Further validation of actigraphy for sleep studies. Sleep. 2003 Feb 1;26(1):81-5. doi: 10.1093/sleep/26.1.81. PMID 12627737
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Brotherton CS, Martin CA, Long MD, Kappelman MD, Sandler RS. Avoidance of Fiber Is Associated With Greater Risk of Crohn's Disease Flare in a 6-Month Period. Clin Gastroenterol Hepatol. 2016 Aug;14(8):1130-6. doi: 10.1016/j.cgh.2015.12.029. Epub 2015 Dec 31. PMID 26748217
- [Background] Voigt RM, Forsyth CB, Green SJ, Mutlu E, Engen P, Vitaterna MH, Turek FW, Keshavarzian A. Circadian disorganization alters intestinal microbiota. PLoS One. 2014 May 21;9(5):e97500. doi: 10.1371/journal.pone.0097500. eCollection 2014. PMID 24848969
- See also: Randomised clinical trial: Deep remission in biologic and immunomodulator naïve patients with crohn's disease - a SONIC post hoc analysis. - PubMed - NCBI [homepage on the Internet]. [cited 6/9/2016]. — https://www.ncbi.nlm.nih.gov/pubmed/25728587

DOCUMENTS (1):
  • Informed Consent Form (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT04637399/ICF_000.pdf